CLINICAL TRIAL: NCT01476969
Title: Effect of Remote Ischemic Perconditioning on Acute Kidney Injury in Adult Valve Replace
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Central South University (Other)
Responsible Party: Principal Investigator, Luo Wanjun, Director, Central South University
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: CentralSouthU
Record Dates: First submitted 2011-11-16; First posted 2011-11-22 (Estimated); Last update posted 2012-08-14 (Estimated); Status verified 2012-08

CONDITIONS: Rheumatic Disease of Heart Valve; Ischemic Reperfusion Injury
Keywords: Ischemia reperfusion injury; Cardiopulmonary bypass; Remote Ischemic Postconditioning; Other Functional Disturbances Following Cardiac Surgery
MeSH Terms: conditions — Reperfusion Injury

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Manual Tourniquet (Experimental)
  Interventions: Device: Remote ischemic postconditioning

INTERVENTIONS:
Device: Remote ischemic postconditioning — the treatment group consisted of three 4-minute cycles left lower limb ischemia,induced by inflating a blood pressure cuff on the lower limb to 600 mmHg with an intervening 4 minutes of reperfusion ,during which time the cuff was deflate;the control group consisted of placing an uninflated cuff on the left lower limb for 24 minutes.The postconditioning protocol was applied after the aortic cross-clamping.
  Other Names: Manual Tourniquet YZ-01

SUMMARY:
The purpose of this study is to determine whether Remote Ischemic Perconditioning is effective on Acute kidney injury in adult valve replacement.

DETAILED DESCRIPTION:
Methods: Patients meeting the requirement will be randomized into 2 groups: the treatment group consisted of three 5-minute cycles left lower limb ischemia, induced by inflating a blood pressure cuff on the lower limb to 600 mmHg with an intervening 5 minutes of reperfusion, during which time the cuff was deflate; the control group consisted of placing an uninflated cuff on the left lower limb for 30 minutes. The postconditioning protocol was applied after the aortic cross-clamping. The clinical data of inotropes requirement, drainage, ventilation and intensive care time will be recorded. Venous blood samples will be taken perioperatively for detecting concentration of troponin I (cTnI), Myocardial enzyme, Renal function, Cystatin c, and High-sensitivity c-reactive protein(HS-CRP).

ELIGIBILITY:
Inclusion Criteria:

* rheumatic heart valve disease requiring selective aortic or double valve(aortic and mitral valve) replacement

Exclusion Criteria:

* infective endocarditis congenital valve disease previous cardiac surgery complicated with rereplace valve
* Renal dysfunction
* diabetes
* coronary artery disease
* hypertension
* peripheral vascular disease affecting the lower limb free of arteriovenous fistula
* receiving aspirin, corticosteroids, angiotensin-converting enzyme inhibitors or statin perioperatively

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2011-09; Primary Completion 2012-11 (Estimated); Study Completion 2012-11 (Estimated)

PRIMARY OUTCOMES:
Renal function | within the first 48h after cardiac surgery

SECONDARY OUTCOMES:
concentration of troponin I (cTnI) | within 48h after cardiac surgery
Myocardial enzyme | within 48h after cardiac surgery
Cystatin C | within 48h after cardiac surgery
High-sensitivity c-reactive protein(HS-CRP) | within 48h after cardiac surgery

CONTACTS AND LOCATIONS:
Overall Officials: Luo Wanjun, M.D., Study Director — Central South University
Locations (1):
- Central South University, Changsha, Hunan, China